CLINICAL TRIAL: NCT04716270
Title: Ablation of Supraventricular Arrhythmias With As Low As Reasonably Achievable X-Ray Exposure (AALARA)
Brief Title: Ablation of Supraventricular Arrhythmias With As Low As Reasonably Achievable X-Ray Exposure
Acronym: AALARA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mohamed Bin Khalifa Bin Sulman Al Khalifa Cardiac Centre (Other Government)
Responsible Party: Sponsor
Other Study IDs: Version 1.0 of 2020-08-05
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Tachycardia, Supraventricular
Keywords: Supraventricular tachycardia; Radiation exposure
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Electrophysiology Study and Ablation — Electrophysiology Study and Ablation of Supraventricular Arrhythmias

SUMMARY:
Observational study is to demonstrate a clinically significant reduction of ionizing radiation exposure during transcatheter ablation of supraventricular tachycardias using the EnSite precision mapping system in a real-world clinical setting without compromising efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patient indicated for supraventricular arrhythmias ablation according to the current guidelines
* Patient is willing to provide written informed consent.

Exclusion Criteria:

* Patient is pregnant.
* Contraindications to ionizing radiation exposure
* Patient's life expectancy is less than 1 year
* Associated complex congenital heart disease
* Cardiac implantable electric devices
* Known pathological venous access to the heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients ≥ 18 years of age, indicated for supraventricular arrhythmias ablation according to the current local applicable guidelines
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure dose | The day of performing the procedure
  The dose of ionizing radiation exposure in patients undergoing Supraventricular Tachycardia catheter ablation utilizing a non-fluoroscopic EnSite Precision 3D mapping system
Incidence of procedure related cardiac Adverse Events (Safety) | 6 months
  Cardiac related serious adverse events frequency during and after ablation procedure of supraventricular arrhythmias

SECONDARY OUTCOMES:
Fluoroscopy time | The day of performing the procedure
  Fluoroscopy time during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Amin, MRCP(UK)FHRS, Principal Investigator — Mohamed Bin Khalifa Cardiac Center
Locations (1):
- Mohamed Bin Khalifa Cardiac Center, Riffa, Bahrain

REFERENCES:
- [Derived] Amin M, Abdrakhmanov A, Kropotkin E, Traykov V, Sallo Z, Geller L, Lorgat F, Sapelnikov O, Toman O, Al-Muti K, Aljaabari M, Bystriansky A, Kornyei L, Mujovic N, Simons S, Szegedi N. Ablation of Supraventricular Arrhythmias With as Low as Reasonably Achievable X-Ray exposure (AALARA): Results of Prospective, Observational, Multicenter, Multinational, Open-Label Registry Study on Real World Data Using Routine Ensite 3D Mapping During SVT Ablation. Pacing Clin Electrophysiol. 2024 Nov;47(11):1441-1448. doi: 10.1111/pace.15075. Epub 2024 Sep 27. PMID 39331462
- [Derived] Szegedi N, Kroptkin E, Traykoc V, Abdrakhmanov A, Lorgat F, Sapelnikov O, Simons S, Amin M. Routine use of a 3D mapping system in the ablation of supraventricular arrhythmias with as low as reasonably achievable X-ray exposure (AALARA): protocol for a prospective, observational, multicentre, multinational, open-label registry study. BMJ Open. 2023 Aug 4;13(8):e072181. doi: 10.1136/bmjopen-2023-072181. PMID 37541748